CLINICAL TRIAL: NCT05225467
Title: Development of Ketoacidosis During the Perioperative Period: an Observational Study 'The DKAP Study'
Acronym: DKAP
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Lars Ivar Pieter Snel, Clinical Research Physician, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: DKAP2022
Record Dates: First submitted 2022-01-05; First posted 2022-02-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ketosis; Keto Acidosis; Ketoses, Metabolic; Ketosis, Diabetic; Peri-operative; Diabetes Mellitus
Keywords: Surgery; Ketones
MeSH Terms: conditions — Ketosis; Diabetic Ketoacidosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: All participants taking part in this study are subsequently categorized in this group

SUMMARY:
Rationale:

During perioperative period, prolonged starvation, surgical stress, acute complications (e.g. infection) and medication changes all promote ketone generation, therefore increasing the risk of ketoacidosis. At present, there is no literature concerning the ketone production in patients undergoing cardiac surgery, regardless of the diabetes status.

Objectives:

The objectives of this study are to explore the change in blood ketone level during the perioperative period in patients with and without diabetes, to observe the incidence of perioperative ketoacidosis, and to investigate therapy and outcome of patients with perioperative ketoacidosis.

DETAILED DESCRIPTION:
Study procedures On the first day of admission, all the patients scheduled for cardiac surgery with an on-pump procedure will be asked for a consent for anonymous using of their information. Patients giving permission will be screened for participation in this study, and those fulfil the inclusion/exclusion criteria will be included for further research.

Blood ketone will be measured with StatStrip Glucose/Ketone Meters (Nova biomedical, United Kingdom) using sample leftover from blood gas analysis. No extra blood draw is needed. The levels of ketones will be measured at four time points:

1. Beginning of surgery;
2. The moment the cardio-pulmonary bypass machine takes over the circulation.
3. After the decoupling of the Cardio-pulmonary bypass machine
4. At the end of surgery.

Diagnosis of ketoacidosis is based on criteria mentioned. Epidemiology characteristics and perioperative variables will be extracted from electronic medical records.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Inclusion Criteria

* Aged eighteen years or older
* Scheduled for open heart surgery

Exclusion criteria

* Diagnosed with type 1 diabetes mellitus or latent auto-immune diabetes in adults
* Recently used sodium glucose transport co-enzyme 2 (SGLT-2i's) within 2 weeks before surgery)
* History of recurrent ketoacidosis (two times or more within three months)
* Emergency surgery
* (Suspected) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery with an on-pump procedure are eligible for inclusion. A total of 54 subjects will be enrolled.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Blood ketone difference | During surgery
  The primary outcome in this study is the difference in blood ketone level before and after cardiac surgery.

SECONDARY OUTCOMES:
Incidence of ketoacidosis | Post surgery up to three days
  The diagnosis criteria for Ketoacidosis are: 1) Beta-hydroxybutyrate (BHB) ≥3 mmol/L or significant ketonuria (≥ ++); 2) blood glucose over 11 mmol/L; and 3) bicarbonate below 15 mmol or arterial potential of hydrogen(pH) less than 7.3.
Difference in ketone development between patient with and without diabetes mellitus. | During Surgery
  Glucose management is compared between two groups to see if there is a potential difference.

OTHER OUTCOMES:
Other | Post surgery up to three days
  Incidence of hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, dr, Principal Investigator — Amsterdam Univeristy medical Center
Locations (1):
- Amsterdam University Medical Centre, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vetter TR, Jones KA. Perioperative Surgical Home: Perspective II. Anesthesiol Clin. 2015 Dec;33(4):771-84. doi: 10.1016/j.anclin.2015.07.002. PMID 26610629
- [Background] Meyer EJ, Mignone E, Hade A, Thiruvenkatarajan V, Bryant RV, Jesudason D. Periprocedural Euglycemic Diabetic Ketoacidosis Associated With Sodium-Glucose Cotransporter 2 Inhibitor Therapy During Colonoscopy. Diabetes Care. 2020 Nov;43(11):e181-e184. doi: 10.2337/dc20-1244. Epub 2020 Sep 17. No abstract available. PMID 32943440
- [Background] Anderson JC, Mattar SG, Greenway FL, Lindquist RJ. Measuring ketone bodies for the monitoring of pathologic and therapeutic ketosis. Obes Sci Pract. 2021 May 4;7(5):646-656. doi: 10.1002/osp4.516. eCollection 2021 Oct. PMID 34631141
- [Background] Thiruvenkatarajan V, Meyer EJ, Nanjappa N, Van Wijk RM, Jesudason D. Perioperative diabetic ketoacidosis associated with sodium-glucose co-transporter-2 inhibitors: a systematic review. Br J Anaesth. 2019 Jul;123(1):27-36. doi: 10.1016/j.bja.2019.03.028. Epub 2019 May 3. PMID 31060732
- [Background] Blanco JC, Khatri A, Kifayat A, Cho R, Aronow WS. Starvation Ketoacidosis due to the Ketogenic Diet and Prolonged Fasting - A Possibly Dangerous Diet Trend. Am J Case Rep. 2019 Nov 22;20:1728-1731. doi: 10.12659/AJCR.917226. PMID 31756175
- [Background] Dennhardt N, Beck C, Huber D, Sander B, Boehne M, Boethig D, Leffler A, Sumpelmann R. Optimized preoperative fasting times decrease ketone body concentration and stabilize mean arterial blood pressure during induction of anesthesia in children younger than 36 months: a prospective observational cohort study. Paediatr Anaesth. 2016 Aug;26(8):838-43. doi: 10.1111/pan.12943. Epub 2016 Jun 13. PMID 27291355
- [Background] Ohkawa H, Iwakawa T, Ohtomo N, Kitayama M, Miyahara A, Ishihara H, Matsuki A. [Clinical study on intraoperative hyperketonemia in non-diabetic surgical patients under general anesthesia]. Masui. 1993 Dec;42(12):1803-7. Japanese. PMID 8301829
- [Background] Polidori D, Iijima H, Goda M, Maruyama N, Inagaki N, Crawford PA. Intra- and inter-subject variability for increases in serum ketone bodies in patients with type 2 diabetes treated with the sodium glucose co-transporter 2 inhibitor canagliflozin. Diabetes Obes Metab. 2018 May;20(5):1321-1326. doi: 10.1111/dom.13224. Epub 2018 Feb 14. PMID 29341404